CLINICAL TRIAL: NCT06652074
Title: Prevalence and Severity of Depression, Anxiety and Stress in a Sample of Resident Doctors in Upper Egypt.
Brief Title: Depression, Anxiety, and Stress in a Sample of Resident Doctors in Upper Egypt
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Sadek Mohamed Megahed, Principal investigator, Assiut University
Other Study IDs: Depression, Anxiety and stress
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the prevalence and severity of symptoms related to depression, anxiety, and stress, among population of resident doctors in Upper Egypt in Assiut University Hospitals and other hospitals in upper Egypt

DETAILED DESCRIPTION:
Many resident doctors during their training experience different levels of stress and this continuous pressure can cause feelings of discouragement and dissatisfaction, which might lead to the desire of leaving a training program.

This pressure could be accompanied by anxiety and depression and have negative effects on clinical performance and even increase the risk of burnout. Adjusting to these hectic job burdens affects individual emotional and intellectual contingency, and the capacity to create a healthy home-work balance. Burnout in residents can have serious effects not only on personal well-being, interpersonal relationships as well as on career but also may have negative effects on patient care .

The prevalence and impact of mental health issues among resident doctors have garnered increasing attention in recent years. Studies suggest that residency training can exacerbate existing vulnerabilities and contribute to the development of mental health disorders. The implications of these conditions are profound, affecting not only the personal well-being of the doctors but also their professional performance, patient care quality, and overall healthcare system efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Resident doctors undergoing post-graduation training in Hospital.
* Resident in hospitals in Upper Egypt

Exclusion Criteria:

* Resident doctors who were already under treatment for any psychiatric disorder and chronic medical illnesses.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: resident doctors in Upper Egypt over age of 20
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-10-10 (Estimated); Study Completion 2026-11-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of symptoms related to depression, anxiety,and stress | 2 years
  To assess the prevalence of symptoms related to depression, anxiety, and stress, among population of resident doctors in Upper Egypt in Assiut University Hospitals and other hospitals in upper Egypt by using the Depression, Anxiety and Stress Scale - 21 (DASS-21)

SECONDARY OUTCOMES:
Severity of symptoms related to depression, anxiety,and stress | 2 years
  To assess the severity of symptoms related to depression, anxiety,and stress by using the Depression, Anxiety and Stress Scale - 21 (DASS-21)

REFERENCES:
- [Background] Meghrajani VR, Marathe M, Sharma R, Potdukhe A, Wanjari MB, Taksande AB. A Comprehensive Analysis of Mental Health Problems in India and the Role of Mental Asylums. Cureus. 2023 Jul 27;15(7):e42559. doi: 10.7759/cureus.42559. eCollection 2023 Jul. PMID 37637646
- [Background] Naji L, Singh B, Shah A, Naji F, Dennis B, Kavanagh O, Banfield L, Alyass A, Razak F, Samaan Z, Profetto J, Thabane L, Sohani ZN. Global prevalence of burnout among postgraduate medical trainees: a systematic review and meta-regression. CMAJ Open. 2021 Mar 8;9(1):E189-E200. doi: 10.9778/cmajo.20200068. Print 2021 Jan-Mar. PMID 33688027
- [Background] Farhangi P, Khajehnasiri F. The prevalence of depression, anxiety, and stress among medical residents: A cross-sectional study in Iran. Acta Medica Iranica. 2020 Nov 19:452-5.